CLINICAL TRIAL: NCT00029731
Title: Arginine Therapy for Acute Chest Syndrome in Sickle Cell Disease
Brief Title: Arginine Treatment of Acute Chest Syndrome (Pneumonia) in Sickle Cell Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FD-R-1978-01; FD-R-001978-01
Record Dates: First submitted 2002-01-21; First posted 2002-01-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Anemia, Sickle Cell; Pneumonia
Keywords: Nitric Oxide; Administration, Oral
MeSH Terms: conditions — Anemia, Sickle Cell; Pneumonia | interventions — Arginine

INTERVENTIONS:
Drug: Arginine hydrochloride

SUMMARY:
This is a study to determine if oral arginine will increase nitric oxide in sickle cell disease (SCD) patients with acute chest syndrome (ACS). It will also assess the effects of arginine in the body and how the body uses nitric oxide in ACS.

DETAILED DESCRIPTION:
Pneumonia in patients with SCD can be particularly severe and has come to be called acute chest syndrome. ACS is a common cause of morbidity in SCD patients and is the most common cause of death in SCD. Multiple factors are involved in the severity of acute pulmonary injury in SCD. Nitric oxide has a multitude of related functions, many of which could impact favorably on ACS in SCD. Nitric oxide is an important inflammatory mediator which is produced by the conversion of L-arginine to citrulline by nitric oxide synthase. Nitric oxide and its precursor, arginine, are known to be low in SCD patients with ACS, suggesting that therapies, such as arginine, aimed at increasing nitric oxide production will improve the clinical course of ACS. Patients will receive 1 of 3 doses of arginine hydrochloride orally 3 times a day for 3 days while hospitalized. The efficacy of arginine will be measured by the increase in nitric oxide production and the physiological effects will be assessed.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of sickle cell disease (Hb SS, SC, or Sbeta thalassemia)

Acute chest syndrome with the following:

* New pulmonary infiltrate on chest radiography involving a full segment of the lung and 1 of the following:
* Fever
* Cough, tachypnea, retractions, rales, or wheezing
* Chest pain

Exclusion criteria:

* Inability to take or tolerate oral medications
* Hepatic dysfunction (SGPT greater than 2 times normal)
* Renal dysfunction (creatinine greater than 2 times normal)
* Mental status or neurological changes
* Allergy to arginine
* History of priapism
* Pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-08; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Oakland, Oakland, California, United States